CLINICAL TRIAL: NCT04735510
Title: Novel Use of Restasis (Cyclosporine Ophthalmic Emulsion 0.05%) on Application of PROSE Devices for Management of Patients With Ocular Surface Disease: A Pilot Study
Brief Title: Novel Use of Restasis and PROSE Devices
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: study redesigned
Sponsor: Boston Sight (Other)
Responsible Party: Principal Investigator, Daniel C Brocks, Principal Investigator, Boston Sight
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFS-RGN-01
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Ocular Surface Disease

STUDY DESIGN:
Intervention Model Description: All participants will receive study drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): This is a single arm study in which all subjects will receive study medication.
  Interventions: Drug: cyclosporine ophthalmic emulsion 0.05%

INTERVENTIONS:
Drug: cyclosporine ophthalmic emulsion 0.05% — All subjects will receive restasis

SUMMARY:
The goal of this prospective observational pilot study is to evaluate the tolerability and safety of RESTASIS (cyclosporine ophthalmic solution 0.05%) when added to the PROSE (Prosthetic Replacement of the Ocular Surface Ecosystem) lens reservoir in patients with ocular surface disease (OSD).

DETAILED DESCRIPTION:
For this study, all subjects will receive Restasis (Cyclosporine ophthalmic emulsion 0.05%). One drop of the dispensed study drop will be instilled in the PROSE lens reservoir twice a day and the remainder of the reservoir will be filled with normal saline (0.9% sodium chloride solution). In order to standardize solutions used in the PROSE reservoir, all patients recruited will be either currently using or will be switched to buffered preservative-free normal saline (Purilens, Lifestyle Inc., pH 7.4 ) to better match the reported pH of RESTASIS (pH 6.5-8.05).

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent has been obtained prior to any study-related procedures taking place
2. Subject is Male or Female, 18 years of age or older prior to the initial visit
3. Is an established wearer of PROSE devices for > 6 months in both eyes
4. Has a finalized PROSE lens design in both eyes, in the opinion of the clinician
5. The PROSE design does NOT include fenestrations
6. Subject requires PROSE devices to treat symptoms and/or signs from underlying dry eye disease, GVHD, Sjogren's syndrome, limbal stem cell deficiency, keratoconjunctivitis sicca, or ocular surface disease
7. Baseline Corneal staining grade of 2 or higher in total, both eyes combined (NEI Grading System)
8. Baseline Ocular Surface Disease Index 13 or greater
9. In the opinion of the investigator, the subject can follow study instructions
10. In the opinion of the investigator, the subject can complete all study procedures and visits
11. Able to wear PROSE device continuously for at least 6 hours at a time without removal, in each eye
12. Able to wear PROSE device for at least 10 total hours a day, in each eye
13. Able to wear PROSE device in subsequent continuous sessions of 6 hours, followed by a break to re-instill Restasis in device bowl, followed by another period of continuous wear of at least 4 hours
14. Currently using buffered preservative free normal saline (Purilens) in the device bowl or willing to transition to buffered preservative free normal saline (Purilens) use in the device bowl during the study

Exclusion Criteria:

1. Is currently participating in any other type of eye-related clinical or research study
2. Is pregnant or nursing as reported by the subject.
3. Has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study.
4. Has had previous ocular surgery within the past 12 weeks.
5. Currently uses or has a prior history of using Restasis in the last 3 months
6. Currently uses or has a prior history of using Cequa in the last 3 months
7. Is currently using Xiidra and has been using Xiidra for less than 3 months
8. Has a history of an allergic reaction or hypersensitivity to any active or inactive ingredient found in Restasis or Cequa or Purilens.
9. Is wearing a PROSE device with Tangible HydraPEG coating
10. The subject is not wearing their PROSE devices daily
11. The subject is only wearing a device for one eye.
12. The participant is monocular
13. The subject wears a PROSE lens with fenestrations
14. The participant carries a diagnosis of glaucoma or ocular hypertension or glaucoma suspect AND is currently using glaucoma medications
15. The participant is NOT able to wear PROSE devices for 6 hours continuously, followed by a break to re-instill Restasis, followed by an additional period of at least 4 hours of continuous wear
16. Allergy to sodium fluorescein
17. Allergy to lissamine green
18. Allergy or intolerance to Purilens solution.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
subjective responses regarding symptoms | Baseline
  Subjects will be given a baseline tolerability questionnaire Disease Index (OSDI)
subjective responses regarding symptoms | 1 week
  Subjects will be given a baseline tolerability questionnaire Disease Index (OSDI)
subjective responses regarding symptoms | 1 month
  Subjects will be given a baseline tolerability questionnaire Disease Index (OSDI)

SECONDARY OUTCOMES:
Oculus keratograph scan | Baseline
  A scan of the eye surface will classify eye redness
Oculus keratograph scan | 1 week
  A scan of the eye surface will classify eye redness
Oculus keratograph scan | 1 month
  A scan of the eye surface will classify eye redness

OTHER OUTCOMES:
Slit lamp exam | Baseline
  The PI will perform a slit lamp exam and staining to measure conjunctival redness
Slit lamp exam | 1 week
  The PI will perform a slit lamp exam and staining to measure conjunctival redness
Slit lamp exam | 1 month
  The PI will perform a slit lamp exam and staining to measure conjunctival redness
Corneal Staining | baseline
  The PI will perform a slit lamp exam and staining to measure corneal staining
Corneal Staining | 1 week
  The PI will perform a slit lamp exam and staining to measure corneal staining
Corneal staining | 1 month
  The PI will perform a slit lamp exam and staining to measure corneal staining

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Brocks, MD, Principal Investigator — Chief Medical Officer
Locations (1):
- BostonSight, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD